CLINICAL TRIAL: NCT02058277
Title: An Open-Label, Randomized, 2-Period Crossover Study To Evaluate The Effect Of A Single Dose Of Aprepitant, A Moderate CYP3A Inhibitor On Bosutinib Administered Orally To Healthy Subjects
Brief Title: A Drug Interaction Study Between Bosutinib And Aprepitant In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1871041
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: bosutinib; aprepitant; drug interaction; healthy volunteers; pharmacokinetics; chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib; Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Other): Healthy volunteers taking a single dose of bosutinib and a single dose of bosutinib plus aprepitant in random order
  Interventions: Drug: bosutinib or bosutinib + aprepitant

INTERVENTIONS:
Drug: bosutinib or bosutinib + aprepitant — Single dose of bosutinib (500 mg) or single dose of bosutinib (500 mg) and aprepitant (125 mg)

SUMMARY:
This is an open label, randomized, single dose, one cohort, two sequence, two period crossover study in healthy subjects. The primary objective of the study is to evaluate the effect of a single oral dose of aprepitant on the pharmacokinetic (PK) profile of a single oral dose of bosutinib in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects with an informed consent document signed and dated by the subject.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of non hormonal contraception as outlined in this protocol .
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area under the Concentration-Time Curve (AUC) | 96 hours
  AUC is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption.
Maximum Observed Plasma Concentration (Cmax) | 96 hours
  Cmax is the peak concentration.

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 96 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 96 hours
  Tmax is measure how fast a drug is absorbed
Plasma Decay Half-Life (t1/2) | 96 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | 96 hours
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 96 hours
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, DeLand, Florida, United States

REFERENCES:
- [Derived] Hsyu PH, Pignataro DS, Matschke K. Effect of aprepitant, a moderate CYP3A4 inhibitor, on bosutinib exposure in healthy subjects. Eur J Clin Pharmacol. 2017 Jan;73(1):49-56. doi: 10.1007/s00228-016-2108-z. Epub 2016 Oct 7. PMID 27718000
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1871041&StudyName=A%20Drug%20Interaction%20Study%20Between%20Bosutinib%20And%20Aprepitant%20In%20Healthy%20Volunteers